CLINICAL TRIAL: NCT04159142
Title: Clinical Study of Nab-paclitaxel Plus Carboplatin Versus Nab-paclitaxel Plus Capecitabine in the Treatment of Advanced Triple-negative Breast Cancer
Brief Title: Nab-paclitaxel Plus Carboplatin Versus Nab-paclitaxel Plus Capecitabine in the Treatment of Advanced Triple-negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Collaborators: Beijing 302 Hospital (Other); CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Cuizhi GENG, Principal Investigator, Hebei Medical University Fourth Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-KAL-BC-16
Record Dates: First submitted 2019-10-23; First posted 2019-11-12 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Triple Negative Breast Cancer; Nab-paclitaxel
Keywords: Nab-paclitaxel; Carboplatin; Capecitabine; Triple Negative Breast Cancer; Maintenance therapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Carboplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nab-paclitaxel + Carboplatin (Experimental): Nab-paclitaxel given IV at 125 mg/m^2 on days 1, 8 and carboplatin given IV at AUC 5 on days 1 every 21 days x 6 cycles； Maintenance therapy: Capecitabine 1000 mg/m^2 bid, d1-14; every 21 days, until disease progression or intolerable toxicity;
  Interventions: Drug: Nab-paclitaxel + Carboplatin
- Nab-paclitaxel + Capecitabine (Experimental): Nab-paclitaxel given IV at 125 mg/m^2 on days 1, 8 and capecitabine given IV at 1000 mg/m^2 bid, d1-14 every 21 days x 6 cycles； Maintenance therapy: Capecitabine 1000 mg/m^2 bid, d1-14; every 21 days, until disease progression or intolerable toxicity;
  Interventions: Drug: Nab-paclitaxel + Capecitabine

INTERVENTIONS:
Drug: Nab-paclitaxel + Carboplatin — nab-paclitaxel given IV at 125 mg/m^2 on days 1, 8 and carboplatin given IV at AUC 5 on days 1 every 21 days x 6 cycles；
  Arms: Nab-paclitaxel + Carboplatin
Drug: Nab-paclitaxel + Capecitabine — Nab-paclitaxel given IV at 125 mg/m^2 on days 1, 8 and capecitabine given IV at 1000 mg/m^2 bid, d1-14 every 21 days x 6 cycles；
  Arms: Nab-paclitaxel + Capecitabine

SUMMARY:
This is a multi-center , open-lable clinical trial. Triple-negative breast cancer (TNBC) is a term applied to breast cancer cases that have <1% expression of the estrogen receptor (ER) and the progesterone receptor (PR) and do not over express HER2. TNBC is diagnosed in 15-20% of breast cancer cases and tends to occur in younger women and have biologically more aggressive high grade disease.

The purpose of this study is to assess the efficacy and safety of the following two combinations: i) nab-paclitaxel+carboplatin; ii) nab-paclitaxel+capecitabine in subjects with advanced TNBC and up to one prior line of systemic treatment for metastatic disease. Maintenance therapy with capecitabine after completion of combination chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Females with age between 18 to 70 years old;
2. Histologically confirmed triple negative breast cancer;
3. No more than one-line prior treatment for locally advanced or metastatic breast cancer;
4. Have at least one measurable lesion as per the RECIST criteria (version 1.1);
5. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to one;
6. Patients with life expectancy of at least 3 months;
7. Bone marrow function：neutrophils (≥1.5×10^9/L), platelets (≥100×10^9/L), hemoglobin (≥90 g/L);
8. Renal and hepatic function: Serum creatinine≤ 1.5×institutional upper limit of normal (ULN); AST and ALT ≤ 2.5 × ULN; Total bilirubin≤1.5×ULN, or patients with Gilbert's syndrome ≤ 2.5 × ULN;
9. Patients had good compliance with the planned treatment, understood the research process and written informed consent.

Exclusion Criteria:

1. Patients with heart disease above grade II (including grade II) identified by New York Heart Association (NYHA) scores;
2. Brain metastasis;
3. Recurrence or metastasis within 6 months after capecitabine withdrawal;
4. Recurrence or metastasis within 6 months after platinum withdrawal;
5. Progression in the treatment, recurrence or metastasis of paclitaxel (including albumin paclitaxel) within 6 months;
6. Patients required clinical intervention with gastrointestinal bleeding, gastrointestinal obstruction and non-feeding;
7. Patients who had Grade 2 or above Peripheral neuropathy;
8. Patients with severe systemic infection or other serious diseases;
9. Patients allergic to or intolerant of chemotherapeutic drugs or their adjuvants;
10. Patients with other malignant tumors in the past five years, except for cured cervical carcinoma in situ and non-melanoma skin cancer;
11. Pregnancy or lactation, as well as reproductive age patients who refused to take appropriate contraceptive measures in the trial;
12. Participation in any trial drug treatment or another interventional clinical trial 30 days before first dose was given;
13. The researchers considered the patients who were not suitable for enrollment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 414 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2028-09-20 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 3 years
  Up to disease progression or death due to any cause

SECONDARY OUTCOMES:
PFS rate for 6 cycles | At the end of Cycle 6 (each cycle is 21 days)
  From the date of randomization to the end of 6 cycles
Objective response rate (ORR) | 3 years
  To evaluate the Overall Response Rate of patients with advanced triple-negative breast cancer
Overall survival (OS) | 3 years
  To evaluate the overall survival of patients with advanced triple-negative breast cancer
Adverse events (AE) | 3 years
  To evaluate the adverse events of patients with advanced triple-negative breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Zefei Jiang, M.D., Study Chair — Beijing 302 Hospital; Cuizhi Geng, M.D., Study Chair — Hebei Medical University Fourth Hospital
Locations (1):
- The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided